CLINICAL TRIAL: NCT01675765
Title: A Phase 1B Study to Evaluate the Safety and Induction of Immune Response of CRS-207 in Combination With Pemetrexed and Cisplatin as Front-line Therapy in Adults With Malignant Pleural Mesothelioma
Brief Title: Safety and Efficacy of Listeria in Combination With Chemotherapy as Front-line Treatment for Malignant Pleural Mesothelioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aduro Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADU-CL-02
Record Dates: First submitted 2012-08-23; First posted 2012-08-30 (Estimated); Results first posted 2020-09-30 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: Cancer; Cancer vaccine; Listeria monocytogenes; Listeria-based vaccines; Pemetrexed; Cisplatin; T regulatory cells; Mesothelin; Malignant Pleural Mesothelioma; Chemotherapy; Standard of care; Naive; Front-line; Immunotherapy; MPM
MeSH Terms: conditions — Mesothelioma, Malignant; Neoplasms | interventions — Immunotherapy; Drug Therapy; Pemetrexed; Cisplatin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immunotherapy plus chemotherapy (Experimental): Weeks 1 and 3: CRS-207 (1 × 10^9 CFU)
  Weeks 5, 8, 11, 14, 17 and 20 (up to 6 cycles every 21 days): pemetrexed (500 mg/m^2) and cisplatin (75 mg/m^2)
  Weeks 23 and 26: CRS-207
  Maintenance Vaccinations: CRS-207 every 8 weeks (starting at Week 34) until disease progression
  Interventions: Biological: Immunotherapy plus chemotherapy
- Immunotherapy with cyclophosphamide plus chemotherapy (Experimental): Weeks 1 and 3: cyclophosphamide (200 mg/m^2), CRS-207 (1 × 10^9 CFU)
  Weeks 5, 8, 11, 14, 17 and 20 (up to 6 cycles every 21 days): pemetrexed (500 mg/m^2) and cisplatin (75 mg/m^2)
  Weeks 23 and 26: cyclophosphamide one day before CRS-207
  Maintenance Vaccinations: cyclophosphamide one day before CRS-207 every 8 weeks (starting at Week 34) until disease progression
  Interventions: Biological: Immunotherapy with cyclophosphamide plus chemotherapy

INTERVENTIONS:
Biological: Immunotherapy plus chemotherapy — live attenuated double deleted Lm
  Other Names: CRS-207; Listeria; pemetrexed; cisplatin; ALIMTA; Platinol
  Arms: Immunotherapy plus chemotherapy
Biological: Immunotherapy with cyclophosphamide plus chemotherapy — live attenuated double deleted Lm
  Other Names: CRS-207; Cytoxan; pemetrexed; cisplatin; ALIMTA; Platinol; Listeria
  Arms: Immunotherapy with cyclophosphamide plus chemotherapy

SUMMARY:
This clinical trial will evaluate the safety and immune response of the sequential administration cancer vaccine CRS-207 (with or without cyclophosphamide) followed by standard of care chemotherapy (pemetrexed and cisplatin). CRS-207 is a weakened (attenuated) form of Listeria monocytogenes that has been genetically-modified to reduce its capacity to cause disease, while maintaining its ability to stimulate potent immune responses. CRS-207 has been engineered to elicit an immune response against the tumor-associated antigen mesothelin, which has been shown to be present at higher levels on certain tumor cells (such as mesothelioma) than on normal cells. Pemetrexed and cisplatin are the standard chemotherapy regimen to treat malignant pleural mesothelioma. This trial will evaluate whether giving CRS-207 cancer vaccine with chemotherapy will induce anti-tumor immune responses and/or objective tumor response.

DETAILED DESCRIPTION:
Up to 60 subjects will be enrolled in this study. Eligible subjects will receive 2 prime vaccinations of CRS-207 (1×10^9 colony-forming units [CFU] given intravenously [i.v.] over 2 hours) (with or without cyclophosphamide) 2 weeks apart followed 2 weeks later by up to 6 cycles of pemetrexed and cisplatin 21 days apart. Three weeks after completion of chemotherapy, subjects will receive an additional 2 infusions (boost vaccinations) of CRS-207 3 weeks apart. Subjects will be followed every 8 weeks until disease progression by immune-related response criteria. Subjects who continue to meet dosing eligibility may receive additional CRS-207 (with or without cyclophosphamide) infusions (maintenance vaccinations) at each follow-up visit.

Study assessments include blood draws for safety and immune response monitoring and CT scans [with optional fluorodeoxyglucose positron emission tomography (FDG-PET)] or magnetic resonance imaging (MRI) to monitor disease status. In addition, optional tumor biopsies may be performed before, during and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically confirmed epithelial or biphasic MPM not amenable to potentially curative surgical resection (subjects with biphasic tumors that have a predominantly (≥50%) sarcomatoid component will be excluded)
* Be at least 18 years of age
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Have an anticipated life expectancy of greater than 6 months
* For women and men of childbearing potential, a medically acceptable method of highly effective contraception (oral hormonal contraceptive, condom plus spermicide, or hormone implants) must be used throughout the study period and for 28 days after their final vaccine administration. (A barrier method of contraception must be employed by all subjects [male and female], regardless of other methods.)
* Be willing and able to give written informed consent, and be able to comply with all study procedures
* Have adequate organ function as defined by specified laboratory values

Exclusion Criteria:

* A candidate for curative surgery
* Surgery within 2 weeks prior to dosing
* Prior radiotherapy or biologic therapy
* Treatment with an investigational agent within 4 weeks before dosing
* Prior systemic chemotherapy
* Currently have or have history of certain study-specified heart, liver, kidney, lung, neurological, immune or other medical conditions
* Documented and ongoing brain metastases
* Have any evidence of hepatic cirrhosis or clinical or radiographic ascites
* Have clinically significant and/or malignant pleural effusion
* Known or suspected allergy or hypersensitivity to yeast or any other component of CRS-207 (e.g., glycerol), Platinol or platinum-containing compounds, or pemetrexed
* Used any systemic steroids within 28 days of study treatment
* Use more than 3 g/d of acetaminophen
* An artificial (prosthetic) joint or other artificial implant or device that cannot be easily removed (with some exceptions for dental and breast implants and biliary stents and mediports)
* Infection with HIV or hepatitis B or C at screening
* Any immunodeficiency disease or immunocompromised state or active autoimmune disease or history of autoimmune disease requiring systemic steroids or other immunosuppressive treatment
* Be a woman who is pregnant or breastfeeding
* Unable to avoid close contact with another individual known to be at high risk of listeriosis (e.g., newborn infant, pregnant woman, HIV-positive individual) during the course of CRS-207 treatment until completion of antibiotic regimen
* Conditions, including alcohol or drug dependence, intercurrent illness, or lack of sufficient peripheral venous access, that would affect the patient's ability to comply with study visits and procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-09-03 (Actual); Primary Completion 2018-09-05 (Actual); Study Completion 2019-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raffit Hassan, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (5):
- United States (5):
  - University of California at San Francisco, San Francisco, California
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - National Cancer Institute, Bethesda, Maryland
  - University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Le DT, Dubenksy TW Jr, Brockstedt DG. Clinical development of Listeria monocytogenes-based immunotherapies. Semin Oncol. 2012 Jun;39(3):311-22. doi: 10.1053/j.seminoncol.2012.02.008. PMID 22595054
- [Derived] Hassan R, Alley E, Kindler H, Antonia S, Jahan T, Honarmand S, Nair N, Whiting CC, Enstrom A, Lemmens E, Tsujikawa T, Kumar S, Choe G, Thomas A, McDougall K, Murphy AL, Jaffee E, Coussens LM, Brockstedt DG. Clinical Response of Live-Attenuated, Listeria monocytogenes Expressing Mesothelin (CRS-207) with Chemotherapy in Patients with Malignant Pleural Mesothelioma. Clin Cancer Res. 2019 Oct 1;25(19):5787-5798. doi: 10.1158/1078-0432.CCR-19-0070. Epub 2019 Jul 1. PMID 31263030

RESULTS

PARTICIPANT FLOW:
Groups:
- Immunotherapy Plus Chemotherapy: Weeks 1 and 3: CRS-207 (1 × 10^9 CFU)
  Weeks 5, 8, 11, 14, 17 and 20 (up to 6 cycles every 21 days): pemetrexed (500 mg/m^2) and cisplatin (75 mg/m^2)
  Weeks 23 and 26: CRS-207
  Maintenance Vaccinations: CRS-207 every 8 weeks (starting at Week 34) until disease progression
  Immunotherapy plus chemotherapy: live attenuated double deleted Lm
- Immunotherapy With Cyclophosphamide Plus Chemotherapy: Weeks 1 and 3: cyclophosphamide (200 mg/m^2), CRS-207 (1 × 10^9 CFU)
  Weeks 5, 8, 11, 14, 17 and 20 (up to 6 cycles every 21 days): pemetrexed (500 mg/m^2) and cisplatin (75 mg/m^2)
  Weeks 23 and 26: cyclophosphamide one day before CRS-207
  Maintenance Vaccinations: cyclophosphamide one day before CRS-207 every 8 weeks (starting at Week 34) until disease progression
  Immunotherapy with cyclophosphamide plus chemotherapy: live attenuated double deleted Lm
Period: Overall Study
Arm/Group | Immunotherapy Plus Chemotherapy | Immunotherapy With Cyclophosphamide Plus Chemotherapy
Started | 38 | 22
Completed | 27 | 14
Not Completed | 11 | 8
Not completed — Progressive disease | 4 | 4
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Death | 1 | 0
Not completed — Clinical progression | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immunotherapy Plus Chemotherapy | Immunotherapy With Cyclophosphamide Plus Chemotherapy | Total
Number analyzed (Participants) | 38 | 22 | 60
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 9 | 6 | 15
  >=65 years | 29 | 16 | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 34 | 17 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 37 | 22 | 59
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 36 | 22 | 58
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 81.63 (16.203) | 73.83 (12.340) | 78.77 (15.271)
Height [Mean (Standard Deviation); unit: cm] | 174.51 (8.295) | 168.41 (7.102) | 172.28 (8.359)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.702 (4.3292) | 26.076 (4.4584) | 26.473 (4.3498)
Body Surface Area [Mean (Standard Deviation); unit: m^2] | 1.982 (0.2230) | 1.852 (0.1756) | 1.935 (0.2148)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Adverse Events
Description: Count of subjects with incidences of adverse events.
Time Frame: From first study dose until 28 days after the final dose (an average of 44 weeks)
Population: Safety Analysis Set (all participants who received >= 1 dose of study treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Immunotherapy Plus Chemotherapy | Immunotherapy With Cyclophosphamide Plus Chemotherapy
Number analyzed (Participants) | 38 | 22
Participants | 38 | 22

2. Primary Outcome: Induction of Immune Response to Mesothelin by Enzyme-linked Immunosorbent Spot (ELISPOT) Assay
Time Frame: Change over time assessed at multiple time points until disease progression or death (up to 12 months or longer)
Population: Immune response to mesothelin was not assessed.
Arm/Group | Immunotherapy Plus Chemotherapy | Immunotherapy With Cyclophosphamide Plus Chemotherapy
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Objective Tumor Response
Description: Objective tumor response was measured using modified Response Evaluation Criteria in Solid Tumors (mRECIST) for assessment of response in malignant pleural mesothelioma (MPM). Per mRECIST for target lesions and assessed by CT: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease, those who fulfilled the criteria for neither PR nor PD; Progressive Disease (PD), >=20% increase in the sum of the longest diameter of target lesions.
Time Frame: Baseline to measured disease progression or death (up to 12 months or longer)
Population: Safety analysis set: all enrolled subjects who received at least one dose of study treatment and had measurable disease.
Measure: Count of Participants; unit: Participants
Arm/Group | Immunotherapy Plus Chemotherapy | Immunotherapy With Cyclophosphamide Plus Chemotherapy
Number analyzed (Participants) | 36 | 21
Participants
  Complete Response | 1 | 0
  Partial Response | 19 | 11
  Stable Disease | 14 | 8
  Progressive Disease | 1 | 2
  Not Assessable | 1 | 0

4. Secondary Outcome: Time to Progression
Time Frame: From date of randomization until date of documented progression (by modified RECIST or immune-related response criteria) or death, assessed up to 12 months or longer
Population: Time to progression was not assessed.
Arm/Group | Immunotherapy Plus Chemotherapy | Immunotherapy With Cyclophosphamide Plus Chemotherapy
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Serum Mesothelin as Correlate of Therapeutic Response
Time Frame: Change over time assessed at multiple time points until disease progression or death (up to 12 months or longer)
Population: Predictive value of serum mesothelin was not assessed.
Arm/Group | Immunotherapy Plus Chemotherapy | Immunotherapy With Cyclophosphamide Plus Chemotherapy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From the start of the first study drug administration until 28 days after the last study drug dose, assessed up to 5 years from the date of randomization.
Arm/Group | Immunotherapy Plus Chemotherapy | Immunotherapy With Cyclophosphamide Plus Chemotherapy
All-Cause Mortality (participants affected / at risk) | 3/38 | 0/22
Serious Adverse Events (participants affected / at risk) | 15/38 | 11/22
Other Adverse Events (participants affected / at risk) | 38/38 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Immunotherapy Plus Chemotherapy (N=38) | Immunotherapy With Cyclophosphamide Plus Chemotherapy (N=22)
Constipation (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chills (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 1
Disease progression (General disorders) | 1 | 0
Influenza like illness (General disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 2
Sepsis (Infections and infestations) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Headache (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Immunotherapy Plus Chemotherapy (N=38) | Immunotherapy With Cyclophosphamide Plus Chemotherapy (N=22)
Chills (General disorders) | 37 | 22
Pyrexia (General disorders) | 37 | 21
Fatigue (General disorders) | 23 | 12
Oedema peripheral (General disorders) | 7 | 3
Non-cardiac chest pain (General disorders) | 5 | 0
Malaise (General disorders) | 3 | 0
Chest pain (General disorders) | 2 | 0
Oedema (General disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 31 | 12
Vomiting (Gastrointestinal disorders) | 25 | 5
Constipation (Gastrointestinal disorders) | 15 | 7
Diarrhoea (Gastrointestinal disorders) | 8 | 2
Abdominal pain (Gastrointestinal disorders) | 4 | 5
Dry mouth (Gastrointestinal disorders) | 4 | 0
Ascites (Gastrointestinal disorders) | 2 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0
Mucosal inflammation (General disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Flatulence (Gastrointestinal disorders) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 19 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 8 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 7 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 4
Dehydration (Metabolism and nutrition disorders) | 5 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 5 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 1
Headache (Nervous system disorders) | 11 | 6
Dizziness (Nervous system disorders) | 8 | 1
Neuropathy peripheral (Nervous system disorders) | 6 | 2
Dysgeusia (Nervous system disorders) | 5 | 0
Syncope (Nervous system disorders) | 2 | 2
Tremor (Nervous system disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Blood creatinine increased (Investigations) | 6 | 7
White blood cell count decreased (Investigations) | 7 | 3
Alanine aminotransferase increased (Investigations) | 7 | 1
Lymphocyte count decreased (Investigations) | 5 | 3
Neutrophil count decreased (Investigations) | 7 | 1
Aspartate aminotransferase increased (Investigations) | 6 | 1
Platelet count decreased (Investigations) | 5 | 2
Weight decreased (Investigations) | 4 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 3
Haemoglobin decreased (Investigations) | 2 | 2
Blood urea increased (Investigations) | 3 | 0
Weight increased (Investigations) | 3 | 0
Blood albumin decreased (Investigations) | 2 | 0
Haematocrit decreased (Investigations) | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 15 | 8
Neutropenia (Blood and lymphatic system disorders) | 3 | 3
Leukopenia (Blood and lymphatic system disorders) | 3 | 0
Leukocytosis (Blood and lymphatic system disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 6 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 5 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Hypotension (Vascular disorders) | 9 | 4
Hypertension (Vascular disorders) | 6 | 2
Flushing (Vascular disorders) | 3 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 0
Jugular vein thrombosis (Vascular disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 4 | 5
Anxiety (Psychiatric disorders) | 1 | 2
Depression (Psychiatric disorders) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 1
Pneumonia (Infections and infestations) | 1 | 2
Sinusitis (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 3 | 0
Sinus tachycardia (Cardiac disorders) | 4 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 2
Tachycardia (Cardiac disorders) | 2 | 1
Tinnitus (Ear and labyrinth disorders) | 5 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 0
Lacrimation increased (Eye disorders) | 6 | 1
Renal impairment (Renal and urinary disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure restriction - study results first published in a joint multi-center paper unless (a) no multi-center publication, or (b) ≥18 months has passed since completion of the study. Thereafter, Investigator may publish provided that Investigator: (i) provides a copy of the publication to Aduro ≥ 30 days in advance of submission for publication; (ii) deletes Aduro Confidential Information (other than the Study results) and (iii) submission may be delayed up to 90 days to permit IP filings."

DOCUMENTS (2):
  • Study Protocol (2018-03-08): https://cdn.clinicaltrials.gov/large-docs/65/NCT01675765/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-04): https://cdn.clinicaltrials.gov/large-docs/65/NCT01675765/SAP_001.pdf